CLINICAL TRIAL: NCT01209104
Title: A Single-dose, Open, Randomized, Crossover Investigation of Age, Gender, Food-effect and Proton-pump Interaction on the Pharmacokinetics of GSK1325756 in Healthy Adult Subjects and a Single-dose, Double Blind, Parallel-group, Placebo- Controlled Investigation of the Pharmacokinetics of GSK1325756
Brief Title: Pharmacokinetics and Safety of GSK1325756 in Elderly Subjects and Adult Subjects of in the Fed and Fasted States and in the Presence of a Proton Pump Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113722
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Nutritional Status
Keywords: omeprazole; proton pump inhibitor; COPD; CXCR2 inhibitor; bioavailability; food-effect
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1-PK and and safety of GSK1325756 in subjects 40-64y (Experimental): This arm assesses the pharmacokinetics and safety of a single oral ose of 100mg of GSK1325756 administered to subjects in the age range 40y-64y when administered in the fasted state, in the presence of a high-fat meal and in the presence of a proton-pump inhibitor.
  Interventions: Drug: GSK1325756
- Cohort 2- PK and safety of GSK1325756 in subjects aged 65y-80y (Experimental): This arm assesses the pharmacokinetics and safety of a single dose of 100mg of GSK1325756 administered to a group of subjects in the 64y-80y age range in the fasted state
  Interventions: Drug: GSK1325756

INTERVENTIONS:
Drug: GSK1325756 — 100mg of a single oral dose of GSK1325756 administered as 2 x 50mg tablets
  Arms: Cohort 1-PK and and safety of GSK1325756 in subjects 40-64y
Drug: GSK1325756 — 100mg of a single oral dose of GSK1325756 administered as 2 x 50mg tablets
  Arms: Cohort 2- PK and safety of GSK1325756 in subjects aged 65y-80y

SUMMARY:
GSK1325756 is a potent, competitive, selective and reversible CXCR2 receptor antagonist that is being developed as a once-daily oral anti-inflammatory medication for the treatment of chronic obstructive pulmonary disease (COPD). Selective antagonism of the interaction between CXCR2 and its various chemokine ligands is a potential strategy for reducing the underlying inflammation in COPD via the inhibition of neutrophil recruitment and activation. The current study explores the effects of age, gender and food (high fat meal) on the pharmacokinetics of GSK1325756.

Because a significant proportion of COPD subjects are prescribed proton pump inhibitors (PPI's) such as omeprazole in order to alleviate symptoms of gastro-esophageal reflux disease (GERD), it is important to understand the absorption of the current formulation of GSK1325756 in an environment of raised intra-gastric pH as will be encountered in patients taking PPI's. Therefore, this study will also evaluate the impact of the proton pump inhibitor omeprazole on the pharmacokinetics of GSK1325756.

DETAILED DESCRIPTION:
GSK1325756 is a potent, competitive, selective and reversible CXCR2 receptor antagonist that is being developed as a once-daily oral anti-inflammatory medication for the treatment of chronic obstructive pulmonary disease (COPD). Selective antagonism of the interaction between CXCR2 and its various chemokine ligands is a potential strategy for reducing the underlying inflammation in COPD via the inhibition of neutrophil recruitment and activation. The current study explores the effects of age, gender and food (high fat meal) on the pharmacokinetics of GSK1325756.

Because a significant proportion of COPD subjects are prescribed proton pump inhibitors (PPI's) such as omeprazole in order to alleviate symptoms of gastro-esophageal reflux disease (GERD), it is important to understand the absorption of the current formulation of GSK1325756 in an environment of raised intra-gastric pH as will be encountered in patients taking PPI's. Therefore, this study will also evaluate the impact of the proton pump inhibitor omeprazole on the pharmacokinetics of GSK1325756.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and study objectives.

   However, subjects taking a stable dose of anti-hypertensive medication for at least 3 months prior to enrollment may be included if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and study objectives. In all cases, subjects should have a resting BP of 140/90 irrespective of anti-hypertensive medication status.

   Subjects taking a stable dose of lipid lowering medications (statins or fibrates) for at least 3 months prior to enrollment may be included if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and study objectives.
2. A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) more than 40 MlU/ml and estradiol less than 40 pg/ml (less than 140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
3. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until least 3-months post-last dose of study drug.
4. Body weight more than or equal to 60 kg (110 lbs) for men and more than or equal to 45 kg (99lbs) for women and BMI within the range 19-32 kg/m2 inclusive.
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
6. Willingness to complete all study procedures and complete all planned treatment periods and follow up assessments.

7.12 lead ECG without any clinically significant abnormality as judged by the Investigator, and average QTcB or QTcF less than 450 msec 8.AST and ALT less than 2xULN; alkaline phosphatase and bilirubin less than 1.5xULN (isolated bilirubin more than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
2. A neutrophil count at screening of less than 2 x 109/L
3. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. A positive pre-study drug/alcohol screen.
5. A positive test for HIV antibody.
6. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of more than 14 drinks for males or more than 7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
9. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures,s compromise subject safety, or interfere with the objectives of the study. All concomitant medications should be queried with the GSK Medical Monitor.
10. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
11. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
12. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
13. Lactating females.
14. Unwillingness or inability to follow the procedures outlined in the protocol.
15. Subject is mentally or legally incapacitated.
16. History of sensitivity to heparin or heparin-induced thrombocytopenia.
17. Urinary cotinine/ exhaled breath CO levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
18. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2010-05-24 (Actual); Study Completion 2010-05-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for GSK1325756 following the administration of a single dose of 100mg of a tablet formulation of GSK1325756 in the fed (after a high-fat meal) and fasted states in healthy adult subjects in the age range 40 to 64 y | 48h of dosing
PK ofGSK1325756 following the administration of a single dose of 100mg of a tablet formulation of GSK1325756 given concomitantly with the final oral dose of 40mg omeprazole on the fifth day of repeat omeprazole dosing in healthy adult subjects 40-64y old | 48h of dosing
PK parameters for GSK1325756 following the administration of a single dose of 100mg of a tablet formulation of GSK1325756 in the fasted state in healthy adult subjects in the age range 65 to 80 years | 48h of dosing

SECONDARY OUTCOMES:
Safety and tolerability of GSK1325756 alone in the fed and fasted states, alone and in combination with 40 mg omeprazole, as assessed by vital signs, ECGs, clinical laboratory data, clinical monitoring, and subject reports of adverse events. | 7-14 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Miller BE, Mistry S, Smart K, Connolly P, Carpenter DC, Cooray H, Bloomer JC, Tal-Singer R, Lazaar AL. The pharmacokinetics and pharmacodynamics of danirixin (GSK1325756)--a selective CXCR2 antagonist --in healthy adult subjects. BMC Pharmacol Toxicol. 2015 Jun 20;16:18. doi: 10.1186/s40360-015-0017-x. PMID 26092545
- See also: Results for study 113722 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113722?search=study&study_ids=113722#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register